CLINICAL TRIAL: NCT07121049
Title: Study on the Influence of Muscle Strength and Physical Fitness Training on Myopia Health Care for Children in Kindergarten
Brief Title: Influence of Strength Training on Myopia Care in Kindergarten Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hungkuang University (Other)
Responsible Party: Principal Investigator, Ciao-Lin Ho, Assistant Professor, Hungkuang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11409
Record Dates: First submitted 2025-07-25; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Myopia; Physical Fitness; Muscle Strength
Keywords: Kindergartens; Muscle training; Myopia
MeSH Terms: conditions — Myopia | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength training group (Experimental): The strength training group participated in 10 weeks of intervention, performing core muscle exercises three times a week between 4 and 6 p.m.
  Interventions: Behavioral: Strength training
- Placebo group (No Intervention): Placebo group did not receive any intervention measures.

INTERVENTIONS:
Behavioral: Strength training — Through systematic muscle training and promotion of outdoor activities, the program integrates early childhood education college students with kindergartens to promote the all-round development of children and establish habits to prevent myopia.
  Arms: Strength training group

SUMMARY:
With the advancement of technology and changes in lifestyle, the physical activity levels of modern children have gradually decreased. This affects their physical health, psychological development, and social skills, and may increase the risk of nearsightedness. Therefore, it is essential to implement muscle training and outdoor activities in schools, travel agencies, and kindergartens. This project aims to promote the comprehensive development of children through systematic muscle training and enhanced outdoor activities, integrating college students from early childhood education programs, travel agencies, and kindergartens to establish habits that prevent nearsightedness.

In the kindergarten setting, 60 children in the senior class will serve as the control group, while another 60 will be in the intervention group. The intervention group will participate in 10 weeks of muscle training and outdoor activities, including core exercises 3 times a week for 60 minutes each session from 4pm to 6pm. Additionally, there will be subsidized a total of 2 outdoor activities on weekends. This approach will not only improve the children's coordination and flexibility but also enhance their physical fitness. Regarding travel agencies, tailored outdoor activities specifically designed for young children can be created, such as ecological explorations and wilderness survival training, allowing children to enjoy the fun of movement and learning in a safe environment. Travel agencies should collaborate with educational institutions to provide professional guidance and safety assurances, giving parents peace of mind. For kindergartens, a comprehensive outdoor activity plan should be established, regularly organizing sports days and group competitions to encourage children to participate in team sports like soccer and relay races. This not only helps improve the children's muscle strength but also fosters their spirit of cooperation and social skills. Through these methods, we aim to effectively increase children's activity levels, promote their overall development, and reduce the risk of nearsightedness.

DETAILED DESCRIPTION:
Body composition includes Metabolic age, body fat percentage, BMI, total body water (%), BMR (Basal Metabolic Rate), Visceral Fat, physique ratings, muscle quality, muscle mass. Body composition was examined by the TANITA RD-545 (Tanita Corporation, Tokyo-Japonya). Tanita Home Page. Available online: https://tanita.eu/understanding-your-measurements (accessed on 13 August 2022). The FSM is a standardized, norm-referenced test of functional strength for children aged 4-10 years (Smits-Engelsman, 2012).

The FSM consists of eight items that measure anaerobic muscular endurance (30-second sit-to-stand times, lateral up-and-down, box lift, and stair test) and muscular strength (overhand throw, underhand throw, chest throw, and standing long jump). For anaerobic muscular endurance items, the number of repetitions in a 30-second period is counted; for muscular strength items, the distance covered is measured in centimeters.

The Visual_Fatigue_Questionnaire is based on the subjective feelings of the subjects and contains 6 questions using a 5-point Likert scale. The subjects are required to circle the score that best describes their current state (1 represents not at all, 2 represents almost not, 3 represents average, 4 represents somewhat severe, and 5 represents very severe) among the following 6 questions.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-7 who are going to be promoted from kindergarten to first grade
* Must be able to exercise

Exclusion Criteria:

* heart disease
* respiratory problems
* severe allergies

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-08-19 (Estimated); Study Completion 2026-08-19 (Estimated)

PRIMARY OUTCOMES:
Change in Spherical Equivalent (SE) | From enrollment to the start of treatment, the end of treatment at 10 weeks
  Mean change in myopia severity. An Independent t-test was conducted to assess the difference in ΔSE (Spherical Equivalent) between the Intervention and Control groups.

SECONDARY OUTCOMES:
Change in Body Fat Percentage | From enrollment to the start of treatment, the end of treatment at 10 weeks
  Body Fat Percentage was examined by the TANITA RD-545 (Tanita Corporation, Tokyo-Japonya). Tanita Home Page. Available online: https://tanita.eu/understanding-your-measurements (accessed on 13 August 2022). A Paired t-test was used to evaluate within-group changes, while an Independent t-test examined the differences between the groups in ΔSE.
Change in FSM Composite Score | From enrollment to the start of treatment, the end of treatment at 10 weeks
  Endurance is determined by the sum of repetitions from the four tests, while strength is measured by the mean distance achieved across the four tests.
Change in Metabolic Age | From enrollment to the start of treatment, the end of treatment at 10 weeks
  Pearson Correlation was utilized to explore the association with ΔSE, while Partial Correlation was calculated while controlling for age. Metabolic age was examined by the TANITA RD-545 (Tanita Corporation, Tokyo-Japonya). Tanita Home Page. Available online: https://tanita.eu/understanding-your-measurements (accessed on 13 August 2022).
Change in Visual Fatigue Score | From enrollment to the start of treatment, the end of treatment at 10 weeks
  Linear Regression analysis was employed, where the ΔScore was modeled as a function of the group and baseline score.
Visceral Fat Responders | From enrollment to the start of treatment, the end of treatment at 10 weeks
  Proportion with ΔVisceral Fat ≤ -10%. A Chi-square test was implemented to determine the differences in responder rates between groups. Visceral Fat was examined by the TANITA RD-545 (Tanita Corporation, Tokyo-Japonya). Tanita Home Page. Available online: https://tanita.eu/understanding-your-measurements (accessed on 13 August 2022).
The correlation between muscle quality and spherical equivalent (SE) | From enrollment to the start of treatment, the end of treatment at 10 weeks
  Bivariate Correlation was analyzed with ΔSE, stratified by group. Muscle Quality was examined by the TANITA RD-545 (Tanita Corporation, Tokyo-Japonya). Tanita Home Page. Available online: https://tanita.eu/understanding-your-measurements (accessed on 13 August 2022).
Hydration-Metabolism Interaction | From enrollment to the start of treatment, the end of treatment at 10 weeks
  A Two-way ANOVA was conducted to assess the effect on ΔSE, considering the interaction between group and hydration tertile.